CLINICAL TRIAL: NCT03006068
Title: A Phase 3 Multicenter, Long-Term Extension Study to Evaluate the Safety and Efficacy of Upadacitinib (ABT-494) in Subjects With Ulcerative Colitis
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of Upadacitinib (ABT-494) in Participants With Ulcerative Colitis (UC)
Acronym: U-ACTIVATE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-533; 2023-505699-31-00 (Other: EU CT)
Record Dates: First submitted 2016-12-20; First posted 2016-12-30 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis (UC); Upadacitinib (ABT-494); Long Term Extension (LTE); Safety; Efficacy; RINVOQ
MeSH Terms: conditions — Colitis, Ulcerative | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Participants receiving Upadacitinib (ABT-494) Dose A (Experimental): The participants in this arm will receive Upadacitinib (ABT-494) dose A.
  Interventions: Drug: Upadacitinib (ABT-494)
- Participants receiving Upadacitinib (ABT-494) Dose B (Experimental): The participants in this arm will receive Upadacitinib (ABT-494) dose B.
  Interventions: Drug: Upadacitinib (ABT-494)
- Participants receiving Upadacitinib (ABT-494) Dose A or Dose B (Experimental): The participants in this arm will receive Upadacitinib (ABT-494) dose A or dose B.
  Interventions: Drug: Upadacitinib (ABT-494)
- Participants receiving Placebo (Experimental): The participants in this arm will receive placebo until study is unblinded.
  Interventions: Drug: Placebo
- Participants receiving Upadacitinib (ABT-494) Dose C (Experimental): The participants in this arm will receive Upadacitinib (ABT-494) dose C.
  Interventions: Drug: Upadacitinib (ABT-494)

INTERVENTIONS:
Drug: Upadacitinib (ABT-494) — Upadacitinib (ABT-494) will be administered orally.
  Other Names: RINVOQ
  Arms: Participants receiving Upadacitinib (ABT-494) Dose A; Participants receiving Upadacitinib (ABT-494) Dose A or Dose B; Participants receiving Upadacitinib (ABT-494) Dose B; Participants receiving Upadacitinib (ABT-494) Dose C
Drug: Placebo — Placebo will be administered orally.
  Arms: Participants receiving Placebo

SUMMARY:
This study is designed to evaluate the long-term safety and efficacy of Upadacitinib in participants with ulcerative colitis (UC) who have not responded at the end of the induction period in Study M14-234 Substudy 1, who have had loss of response during the maintenance period of Study M14-234 Substudy 3, or who have successfully completed Study M14-234 Substudy 3.

ELIGIBILITY:
Inclusion Criteria:

Note: Participants aged 16 or 17 may enroll in M14-234 or M14-675 where locally permissible

* Participant has not achieved clinical response at the end of the induction period (Week 8) in Study M14-234 Substudy 1, has had loss of response during the maintenance period of Study M14-234 Substudy 3, or has successfully completed Study M14-234 Substudy 3. During the COVID-19 pandemic, for participants with missing endoscopy at Week 8, Week 16 or Week 52 due to the COVID-19 pandemic in Studies M14-234 Substudy 2, M14-234 Substudy 3 and M14-675, participants may be enrolled if certain criteria are met.
* If female, participant must meet the contraception criteria.
* Women of childbearing potential must have a negative urine pregnancy test at Week 0 visit.
* Participant is judged to be in otherwise good health as determined by the principal investigator based upon clinical evaluations performed during the preceding study (Study M14-234).
* Must be able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

* For any reason participant is considered by the investigator to be an unsuitable candidate.
* Female participant with a positive pregnancy test at the final visit of Study M14-234 or who is considering becoming pregnant during the study or within 30 days after the last dose of study drug.
* Known hypersensitivity to upadacitinib or its excipients or had any adverse event (AE) during the preceding studies, that in the investigator's judgment makes the participant unsuitable for this study.
* Participant with an active or recurrent infection that based on the investigator's clinical assessment makes the participant an unsuitable candidate for the study. Participants with ongoing infections undergoing treatment may be enrolled BUT NOT dosed until the infection has been successfully treated.
* Current evidence of active tuberculosis (TB); current evidence of latent tuberculosis and for any reason the participant cannot take full course of TB prophylaxis treatment as required per protocol.
* Participant with a poorly controlled medical condition, such as uncontrolled diabetes, unstable ischemic heart disease, moderate or severe congestive heart failure (New York Heart Association class III or IV), recent cerebrovascular accidents and any other condition which, in the opinion of the investigator or sponsor, would put the subject at risk by participation in this study.
* Participants have malignancy, high-grade dysplasia, un-removed low-grade dysplasia of the gastrointestinal tract diagnosed at the endoscopy performed at the final visit of Study M14-234.
* History of any malignancy except for successfully treated nonmelanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix from evaluations performed in Study M14-234.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessing Treatment-Emergent Adverse Events | Up to 288 Weeks
  Treatment-emergent adverse events are defined as events that begin or worsen either on or after the first dose of the study drug and within 30 days after the last dose of the study drug in the analysis period.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (492):
- United States (147):
  - East View Medical Research, LLC /ID# 171184, Mobile, Alabama
  - CB Flock Research Corporation /ID# 165986, Mobile, Alabama
  - Delsol Research Management, Ll /Id# 170130, Chandler, Arizona
  - Digestive Disease Consultants, A Division of Arizona Digestive Health, P.C /ID# 211886, Mesa, Arizona
  - Duplicate_Arizona Arthritis & Rheumatology Research, PLLC /ID# 169823, Sun City, Arizona
  - Adobe Clinical Research LLC /ID# 155249, Tucson, Arizona
  - Duplicate_University of Arizona /ID# 150568, Tucson, Arizona
  - Citrus Valley Gastroenterology /ID# 151915, Covina, California
  - Newport Huntington Medical Group /ID# 217006, Huntington Beach, California
  - UC San Diego Health System /ID# 155187, La Jolla, California
  - United Medical Doctors /ID# 207467, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 216830, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 157082, Los Angeles, California
  - Facey Medical Foundation /ID# 203135, Mission Hills, California
  - United Medical Doctors - Murrieta /ID# 151213, Murrieta, California
  - Ventura County Gastroenterology Medical Group /ID# 163417, Oxnard, California
  - Inland Empire Clinical Trials, LLC /ID# 216163, Rialto, California
  - San Diego Clinical Trials /ID# 212121, San Diego, California
  - Medical Assoc Research Grp /ID# 169149, San Diego, California
  - Univ of California San Francis /ID# 164583, San Francisco, California
  - Delta Waves, Inc. /ID# 151727, Colorado Springs, Colorado
  - South Denver Gastroenterology /ID# 151224, Lone Tree, Colorado
  - Western States Clinical Res /ID# 158078, Wheat Ridge, Colorado
  - Duplicate_Western Connecticut Medical Group /ID# 169211, Danbury, Connecticut
  - Gastroenterology Center of Connecticut /ID# 150534, Hamden, Connecticut
  - West Central Gastroenterology /ID# 155242, Clearwater, Florida
  - Moonshine Research Center, Inc /ID# 152534, Doral, Florida
  - Universal Axon Clinical Research /ID# 213463, Doral, Florida
  - Palmetto Research, LLC /ID# 151724, Hialeah, Florida
  - Nature Coast Clinical Research - Inverness /ID# 154070, Inverness, Florida
  - Encore Borland-Groover Clinical Research /Id# 170913, Jacksonville, Florida
  - SIH Research Mumtaz, Inc /ID# 163199, Kissimmee, Florida
  - Cfagi Llc /Id# 202018, Maitland, Florida
  - Duplicate_University of Miami /ID# 215443, Miami, Florida
  - Advanced Pharma CR, LLC /ID# 151723, Miami, Florida
  - New Horizon Research Center /ID# 152475, Miami, Florida
  - Crystal Pharmacology Research /ID# 151848, Miami, Florida
  - Coral Research Clinic /ID# 150524, Miami, Florida
  - Advanced Research Institute, Inc /ID# 163093, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 151725, Orlando, Florida
  - Omega Research Group /ID# 200271, Orlando, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 201791, Tampa, Florida
  - Duplicate_University of South Florida /ID# 214494, Tampa, Florida
  - Duplicate_AdventHealth Tampa /ID# 200274, Tampa, Florida
  - Gastroenterology Associates of Central Georgia, LLC /ID# 165783, Macon, Georgia
  - Infinite Clinical Trials /ID# 215342, Riverdale, Georgia
  - Atlanta Gastroenterology Spec /ID# 150565, Suwanee, Georgia
  - Next Innovative Clinical Research - Chicago /ID# 217323, Chicago, Illinois
  - Duplicate_The University of Chicago DCAM /ID# 150564, Chicago, Illinois
  - Duplicate_NorthShore University HealthSystem /ID# 150570, Evanston, Illinois
  - Northwest Health Care Associates /ID# 151591, Hoffman Estates, Illinois
  - Carle Foundation Hospital /ID# 151155, Urbana, Illinois
  - MediSphere Medical Research Center /ID# 152080, Evansville, Indiana
  - Indianapolis Gastroenterology /ID# 162914, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics /ID# 157059, Iowa City, Iowa
  - Cotton O'Neil Clinical Research Center, Digestive Health /ID# 167183, Topeka, Kansas
  - Tri-State Gastroenterology /ID# 169812, Crestview Hills, Kentucky
  - Houma Digestive Health Special /ID# 151851, Houma, Louisiana
  - Nola Research Works, LLC /ID# 153365, New Orleans, Louisiana
  - Louisiana Research Center, LLC /ID# 150526, Shreveport, Louisiana
  - University of Maryland, Baltimore /ID# 150529, Baltimore, Maryland
  - Gastro Center of Maryland /ID# 200024, Columbia, Maryland
  - Massachusetts General Hospital /ID# 165678, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 151158, Ann Arbor, Michigan
  - Huron Gastroenterology Assoc /ID# 152712, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 153031, Chesterfield, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 161983, Chesterfield, Michigan
  - Revival Research Institute, LLC /ID# 207281, Southfield, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 157487, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 151681, Rochester, Minnesota
  - Minnesota Gastroenterology PA /ID# 151682, Saint Paul, Minnesota
  - University of Mississippi Medical Center /ID# 213140, Jackson, Mississippi
  - Southern Therapy and Advanced Research (STAR) LLC /ID# 170713, Jackson, Mississippi
  - Washington University-School of Medicine /ID# 150537, St Louis, Missouri
  - Vector Clinical Trials /ID# 153052, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 150566, Lebanon, New Hampshire
  - Cooper Gastroenterology at Fire Road /ID# 153048, Egg Harbor, New Jersey
  - Atlantic Digestive Health Inst /ID# 150527, Morristown, New Jersey
  - Rutgers Robert Wood Johnson /ID# 155247, New Brunswick, New Jersey
  - Duplicate_University of New Mexico Department of Internal Medicine /ID# 214399, Albuquerque, New Mexico
  - NY Scientific /ID# 152708, Brooklyn, New York
  - Duplicate_NYU Langone Long Island Clinical Research Association /ID# 155271, Great Neck, New York
  - Columbia Univ Medical Center /ID# 163409, New York, New York
  - Duplicate_DiGiovanna Institute for Medical Education & Research /ID# 201534, North Massapequa, New York
  - Premier Medical Group - GI Division /ID# 153366, Poughkeepsie, New York
  - Gastoenterology Group of Rochester /ID# 151080, Rochester, New York
  - Richmond University Medical Center /ID# 201860, Staten Island, New York
  - Montefiore Medical Center - Moses Campus /ID# 150559, The Bronx, New York
  - Advantage Clinical Trials /ID# 163940, The Bronx, New York
  - Digestive Health Partners - Biltmore Office /ID# 167238, Asheville, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 157060, Charlotte, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC /ID# 150561, Charlotte, North Carolina
  - Atlantic Gastroenterology Clinical Research /ID# 151901, Greenville, North Carolina
  - Clinical Trials of America /ID# 153453, Winston-Salem, North Carolina
  - Duplicate_Atrium Health Wake Forest Baptist Medical Center /ID# 150528, Winston-Salem, North Carolina
  - Plains Clinical Research Center, LLC /ID# 170291, Fargo, North Dakota
  - Gastro Health Research /ID# 151683, Cincinnati, Ohio
  - University Of Cincinnati Medical Center /ID# 164584, Cincinnati, Ohio
  - The Ohio State University /ID# 169417, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 169697, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 200066, Dayton, Ohio
  - Dayton Gastroenterology, Inc. /ID# 167632, Englewood, Ohio
  - Great Lakes Gastroenterology Research, LLC /ID# 201773, Mentor, Ohio
  - Ohio Clinical Research Partner /ID# 154074, Mentor, Ohio
  - Hightower Clinical /ID# 216338, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 201057, Oklahoma City, Oklahoma
  - Options Health Research, LLC /ID# 150569, Tulsa, Oklahoma
  - Healthcare Research Consultant /ID# 163096, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic /ID# 152528, Portland, Oregon
  - Guthrie Medical Group, PC /ID# 150533, Sayre, Pennsylvania
  - Penn State Health Colonnade /ID# 150267, State College, Pennsylvania
  - Pharmacorp Clinical Trials /ID# 153363, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 150557, Greenville, South Carolina
  - Gastro One /ID# 151154, Cordova, Tennessee
  - Duplicate_East Tennessee Research Institute /ID# 203611, Johnson City, Tennessee
  - Quality Medical Research /ID# 203427, Nashville, Tennessee
  - Vanderbilt University Medical Center /ID# 153364, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 151528, Arlington, Texas
  - Inquest Clinical Research /ID# 164636, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209949, Cedar Park, Texas
  - GI Alliance /ID# 209806, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 200771, Dallas, Texas
  - Digestive Health Associates of Texas (DHAT) Research Institute - Garland /ID# 151221, Garland, Texas
  - Vilo Research Group Inc /ID# 212626, Houston, Texas
  - CliniCore International, LLC /ID# 152078, Houston, Texas
  - Duplicate_Baylor College of Medicine - Baylor Medical Center /ID# 150538, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201217, Houston, Texas
  - GI Specialists of Houston /ID# 202337, Houston, Texas
  - Duplicate_Caprock Gastro Research, LLC /ID# 215116, Lubbock, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 167954, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 169397, San Antonio, Texas
  - Carl R. Meisner Medical Clinic /ID# 171270, Sugar Land, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 204777, Temple, Texas
  - Tyler Research Institute, LLC /ID# 169147, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 167764, Victoria, Texas
  - HP Clinical Research /ID# 163941, Bountiful, Utah
  - Advanced Research Institute /ID# 162640, Ogden, Utah
  - Utah Gastroenternology - St. Mark's Office /ID# 163097, Salt Lake City, Utah
  - Duplicate_Velocity Clinical Research - Salt Lake City /ID# 163180, West Jordan, Utah
  - Ctr for Gastrointestinal Healt /ID# 153369, Franklin, Virginia
  - Texas Digestive Disease Consultants, PLLC dba GI Alliance /ID# 163630, Bellevue, Washington
  - Virginia Mason Hospital & Medical Center /ID# 153030, Seattle, Washington
  - The Polyclinic /ID# 165117, Seattle, Washington
  - The Vancouver Clinic, INC. PS /ID# 162334, Vancouver, Washington
  - Aurora Medical Center - Grafto /ID# 151726, Grafton, Wisconsin
  - Wisconsin Center for Advanced Research /ID# 151845, Milwaukee, Wisconsin
  - Duplicate_Medical College of Wisconsin /ID# 151850, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Britanico de Buenos Aires /ID# 209496, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Cardio Alem /ID# 211281, San Isidro, Buenos Aires
  - Gedyt /ID# 210016, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Mautalen Salud e Investigacion /ID# 171174, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Sanatorio 9 de Julio /ID# 150215, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 164186, Córdoba
- Australia (6):
  - Macquarie University Hospital /ID# 211953, Macquarie University, New South Wales
  - Mater Misericordiae Limited /ID# 212686, South Brisbane, Queensland
  - Griffith University /ID# 211954, Southport, Queensland
  - Monash Health - Monash Medical Centre /ID# 150218, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 152503, Fitzroy Melbourne, Victoria
  - Fiona Stanley Hospital /ID# 211641, Murdoch, Western Australia
- Austria (4):
  - Ordensklinikum Linz GmbH Barmherzige Schwestern /ID# 150462, Linz, Upper Austria
  - Klinik Landstrasse /ID# 162867, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 150616, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 150463, Salzburg
- Vitebsk Regional Advanced Clin /ID# 169592, Vitebsk, Belarus
- Belgium (3):
  - Universitair Ziekenhuis Leuven /ID# 150468, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 150467, Roeselare, West-Vlaanderen
  - AZ Maria Middelares /ID# 150466, Ghent
- Bosnia and Herzegovina (5):
  - Duplicate_University Clinical Centre of the Republic of Srpska /ID# 150223, Banja Luka, Republika Srpska
  - Duplicate_University Clinical Centre of the Republic of Srpska /ID# 150712, Banja Luka, Republika Srpska
  - University Clinical Center Tuzla /ID# 150224, Tuzla, Tuzlanski
  - University Clinical Hospital Mostar /ID# 150711, Mostar
  - Clinical Center University of Sarajevo /ID# 150222, Sarajevo
- Brazil (7):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva /ID# 153744, Goiânia, Goiás
  - Faculdade de Medicina do ABC /ID# 152489, Santo André, La Spezia
  - Hospital Nossa Senhora das Graças /ID# 152488, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre /ID# 153745, Porto Alegre, Rio Grande do Sul
  - Upeclin Fmb - Unesp /Id# 152493, Botucatu, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 152492, Ribeirão Preto, São Paulo
  - Kaiser Clinica e Hospital Dia /ID# 152491, São José do Rio Preto, São Paulo
- Canada (16):
  - University of Calgary /ID# 151818, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 211169, Edmonton, Alberta
  - University of Alberta Hospital /ID# 151824, Edmonton, Alberta
  - Covenant Health /ID# 158931, Edmonton, Alberta
  - OCT Research ULC /ID# 153179, Kelowna, British Columbia
  - Percuro Clinical Research, Ltd /ID# 150479, Victoria, British Columbia
  - Medicor Research Inc /ID# 151825, Greater Sudbury, Ontario
  - Duplicate_Hamilton Health Sciences -McMaster University Medical Centre /ID# 150477, Hamilton, Ontario
  - Ottawa Hospital Research Institute /ID# 151817, Ottawa, Ontario
  - Toronto Digestive Disease Associates /ID# 150475, Vaughan, Ontario
  - CISSS de la Monteregie /ID# 159271, Greenfield Park, Quebec
  - Duplicate_CISSS de Chaudière-Appalaches, Hôpital Hotel-Dieu de Lévis /ID# 150473, Lévis, Quebec
  - Recherche GCP Research /ID# 151819, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CRCHUM /ID# 167170, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre /ID# 170013, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 150478, Sherbrooke, Quebec
- Chile (6):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 212425, Concepción, Bio-Bio
  - CTR Estudios Clinicos /ID# 200111, Providencia, Region Metropolitana Santiago
  - M y F Estudios Clínicos /ID# 200112, Santiago, Region Metropolitana Santiago
  - Centro de Investigaciones Clínicas Viña del Mar /ID# 150226, Viña del Mar, Región de Valparaíso
  - Research Group /ID# 203177, Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad De Los Andes /ID# 207427, Santiago
- China (16):
  - The First Affiliated Hospital, Sun Yat-sen University /ID# 150517, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 150518, Guangzhou, Guangdong
  - Affiliated Taihe Hospital of Hubei University of Medicine /ID# 216407, Shiyan, Hubei
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Techno /ID# 167089, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 167079, Wuhan, Hubei
  - Duplicate_Xiangya Hospital Central South University /ID# 167230, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University /ID# 212185, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 210087, Changchun, Jilin
  - Shengjing Hospital of China Medical University /ID# 166921, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 150523, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital /ID# 150522, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 165826, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 167041, Chengdu, Sichuan
  - Tianjin Medical University General Hospital /ID# 170605, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 165813, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital,Meical School Zhejiang University /ID# 150516, Hangzhou, Zhejiang
- Colombia (3):
  - Hospital Universitario de San /ID# 155388, Medellín, Antioquia
  - Coorp Hosp Juan Ciudad Sede Hospital Universitario Mayor Mederi /ID# 152811, Bogota DC, Cundinamarca
  - Imat Oncomedica /ID# 207052, Montería, Departamento de Córdoba
- Croatia (8):
  - Duplicate_Poliklinika Solmed /ID# 211567, Grad Zagreb, City of Zagreb
  - Klinicka bolnica Dubrava Zagreb /ID# 150228, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 150262, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 150715, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Osijek /ID# 150229, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 150714, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 213989, Split, Split-Dalmatia County
  - Zadar General Hospital /ID# 150261, Zadar
- Czechia (7):
  - Iscare Klinické Centrum /ID# 209279, Prague, Praha 9
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 150946, Hradec Králové
  - CTCenter MaVe s.r.o. /ID# 150903, Olomouc
  - ARTROSCAN s.r.o. /ID# 150502, Ostrava
  - Nemocnice Pardubickeho kraje, a.s. /ID# 213541, Pardubice
  - Nemocnice Milosrdnych sester sv. Karla Boromejskeho v Praze /ID# 216224, Prague
  - Axon Clinical, s.r.o. /ID# 152477, Prague
- Estonia (4):
  - North Estonia Medical Centre /ID# 160871, Mustamäe, Harju
  - West Tallinn Central Hospital /ID# 150490, Tallinn, Harju
  - East Tallinn Central Hospital - Magdaleena Unit /ID# 150488, Tallinn, Harju
  - Tartu University Hospital /ID# 150489, Tartu
- Finland (5):
  - Tampereen yliopistollinen sairaala /ID# 150376, Tampere, Pirkanmaa
  - Turku University Hospital /ID# 169895, Turku, Southwest Finland
  - Duplicate_Helsinki Univ Central Hospital /ID# 154283, Helsinki
  - Keski-Suomen Sairaala Nova /ID# 155665, Jyväskylä
  - Laakarikeskus Ikioma /ID# 150377, Mikkeli
- France (6):
  - Chu de Nice-Hopital Larchet Ii /Id# 152608, Nice, Alpes-Maritimes
  - CHU Montpellier - Hopital Saint Eloi /ID# 200088, Montpellier, Herault
  - CHRU Lille - Hopital Claude Huriez /ID# 152609, Lille, Nord
  - HCL - Hopital Lyon Sud /ID# 152540, Pierre-Bénite, Rhone
  - Centre Hospitalier Departemental Vendee (Chd Vendee) /ID# 165749, La Roche-sur-Yon, Vendee
  - CHU de Saint-Etienne, Hopital Nord /ID# 165756, Saint-Etienne
- Germany (10):
  - Universitatsklinikum Mannheim /ID# 150405, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 151698, Tübingen, Baden-Wurttemberg
  - Duplicate_Agaplesion Markus Krankenhaus /ID# 161870, Frankfurt am Main, Hesse
  - Duplicate_Universitaetsklinikum Muenster /ID# 150402, Munster, Lower Saxony
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 214575, Herne, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 215812, Saarbrücken, Saarland
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 161871, Kiel, Schleswig-Holstein
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 151697, Berlin
  - Medizinisches Versorgungszentrum Portal 10 /ID# 207136, Münster
  - Praxis medicum /ID# 150404, Wiesbaden
- Greece (7):
  - General Hospital of Athens Laiko /ID# 208672, Athens, Attica
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 202101, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 150236, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 150406, Athens
  - University General Hospital of Ioannina /ID# 164247, Ioannina
  - Theageneio Anticancer Hospital /ID# 164187, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 209522, Thessaloniki
- Hungary (6):
  - Meditres Kft. /ID# 151597, Kecskemét, Bács-Kiskun county
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 150410, Szombathely, Vas County
  - Bekes Megyei Kozponti Korhaz /ID# 151601, Békéscsaba
  - Semmelweis Egyetem /ID# 150409, Budapest
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet /ID# 151599, Sopron
  - Mentahaz Maganorvosi Kozpont /ID# 206977, Székesfehérvár
- Ireland (5):
  - St James Hospital /ID# 150413, Dublin, Dublin
  - St Vincents University Hospital /ID# 150411, Elm Park, Dublin
  - Mercy University Hospital /ID# 153794, Cork
  - Beaumont Hospital /ID# 150414, Dublin
  - University Hospital Galway /ID# 150412, Galway
- Israel (4):
  - Shaare Zedek Medical Center /ID# 163139, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 165119, Jerusalem, Jerusalem
  - Soroka University Medical Center /ID# 156562, Beersheba, Southern District
  - Rambam Health Care Campus /ID# 150416, Haifa
- Italy (10):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 150424, Bologna, Emilia-Romagna
  - IRCCS Istituto Clinico Humanitas /ID# 151363, Rozzano, Lombardy
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico /ID# 150605, Milan, Milano
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 216673, Rho, Milano
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 150425, Rome, Roma
  - Duplicate_Azienda Ospedaliera San Camillo Forlanini /ID# 151362, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 150420, Rome, Roma
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 201726, Negrar, Verona
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 150421, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 150263, Palermo
- Japan (74):
  - Aichi Medical University Hospital /ID# 151994, Nagakute, Aichi-ken
  - Nagoya University Hospital /ID# 152728, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 151949, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital /ID# 171470, Toyohashi, Aichi-ken
  - Ieda Hospital /ID# 157782, Toyota-shi, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center /ID# 152761, Hirosaki-shi, Aomori
  - Tokatsu Tsujinaka Hospital /ID# 214964, Abiko-shi, Chiba
  - Tsujinaka Hospital - Kashiwanoha /ID# 209572, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 151935, Sakura-shi, Chiba
  - Juntendo University Urayasu Hospital /ID# 208783, Urayasu-shi, Chiba
  - Fukui Prefectural Hospital /ID# 210450, Fukui-shi, Fukui
  - Fukuoka University Chikushi Hospital /ID# 152627, Chikushino-shi, Fukuoka
  - Saiseikai Fukuoka Genaral Hospital /ID# 209481, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 152525, Fukuoka, Fukuoka
  - Duplicate_Kitakyushu Municipal Medical Center /ID# 152589, Kitakyushu, Fukuoka
  - Kurume University Hospital /ID# 151977, Kurume-shi, Fukuoka
  - Ogaki Municipal Hospital /ID# 208226, Ogaki-shi, Gifu
  - National Hospital Organization Fukuyama Medical Center /ID# 206294, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 151952, Hiroshima, Hiroshima
  - Duplicate_Asahikawa Medical University Hospital /ID# 170281, Asahikawa-shi, Hokkaido
  - Obihiro kosei Hospital /ID# 210425, Obihiro-shi, Hokkaido
  - Sapporo Tokushukai Hospital /ID# 209449, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 151705, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 206493, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 208495, Sapporo, Hokkaido
  - Aoyama Clinic /ID# 152048, Kobe, Hyōgo
  - Duplicate_Hyogo Medical University Hospital /ID# 152433, Nishinomiya-shi, Hyōgo
  - Duplicate_National Hospital Organization Mito Medical Center /ID# 152626, Higashi Ibaraki-gun, Ibaraki
  - Kanazawa University Hospital /ID# 207810, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center /ID# 203412, Morioka, Iwate
  - Imamura General Hospital /ID# 227138, Kagoshima, Kagoshima-ken
  - Idzuro Imamura Hospital /ID# 207640, Kagoshima, Kagoshima-ken
  - Sameshima Hospital /ID# 206673, Kagoshima, Kagoshima-ken
  - Kagoshima IBD Gastroenterology Clinic /ID# 245222, Kagoshima, Kagoshima-ken
  - St Marianna University School Of Medicine /ID# 209452, Kawasaki-shi, Kanagawa
  - SHOWA Medical University Fujigaoka Hospital /ID# 208223, Yokohama, Kanagawa
  - Yokohama City University Medical Center /ID# 169900, Yokohama, Kanagawa
  - Japanese Red Cross Kyoto Daiichi Hosital /ID# 152358, Kyoto, Kyoto
  - Kyoto University Hospital /ID# 211808, Kyoto, Kyoto
  - Mie University Hospital /ID# 207253, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 214349, Yokkaichi-shi, Mie-ken
  - National Hospital Organization Sendai Medical Center /ID# 209529, Sendai, Miyagi
  - NHO Nagasaki Medical Center /ID# 210821, Omura-shi, Nagasaki
  - Kenseikai Dongo Hospital /ID# 208102, Yamatotakada-shi, Nara
  - Saiseikai Niigata Hospital /ID# 209923, Niigata, Niigata
  - Duplicate_Niigata University Medical & Dental Hospital /ID# 218050, Niigata, Niigata
  - Ishida Clinic of IBD and Gastroenterology /ID# 210118, Ōita, Oita Prefecture
  - Chikuba Hospital for Proctological and Gastrointestinal Diseases /ID# 157820, Kurashiki-shi, Okayama-ken
  - Duplicate_Okayama University Hospital /ID# 217924, Okayama, Okayama-ken
  - Kinshukai Infusion Clinic /ID# 207866, Osaka, Osaka
  - Kitano Hospital, Tazuke Kofukai Medical Research Institute /ID# 210396, Osaka, Osaka
  - Osaka City General Hospital /ID# 152703, Osaka, Osaka
  - Osaka Red Cross Hospital /ID# 209477, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 152681, Osaka, Osaka
  - Shoyukai Fujita Gastroenterological Hospital /ID# 216494, Takatsuki-shi, Osaka
  - Toyonaka Municipal Hospital /ID# 217083, Toyonaka-shi, Osaka
  - Duplicate_Saga University Hospital /ID# 209272, Saga, Saga-ken
  - Saitama Medical Center /ID# 152019, Kawagoe, Saitama
  - Tokitokai Tokito clinic /ID# 152676, Saitama-shi, Saitama
  - National Hospital Organization Higashi-Ohmi General Medical Center /ID# 210711, Higashi-ohmi-shi, Shiga
  - Shimane University Hospital /ID# 208906, Izumo-shi, Shimane
  - Hamamatsu University Hospital /ID# 205709, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 163571, Sunto-gun, Shizuoka
  - Institute of Science Tokyo Hospital /ID# 152017, Bunkyo-ku, Tokyo
  - St. Lukes International Hospital /ID# 208075, Chuo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 152584, Hachioji-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 152687, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 153195, Mitaka-shi, Tokyo
  - Duplicate_Center hospital of the National Center for Global Health and Medicine /ID# 209533, Shinjuku-ku, Tokyo
  - Duplicate_Tokyo Women's Medical University Hospital /ID# 205978, Shinjuku-ku, Tokyo
  - Yamagata University Hospital /ID# 171468, Yamagata, Yamagata
  - Tokuyama Central Hospital /ID# 216995, Shunan-shi, Yamaguchi
  - Yamanashi Prefectural Central Hospital /ID# 151909, Kofu, Yamanashi
  - Teikyo University Hospital /ID# 209865, Tokyo
- Latvia (2):
  - VCA Polyclinic Aura /ID# 150436, Riga
  - Pauls Stradins Clinical University Hospital /ID# 153183, Riga
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 150439, Kaunas
  - Klaipeda university hospital /ID# 163501, Klaipėda
  - Klaipeda University Hospital /ID# 163719, Klaipėda
  - Duplicate_Vilnius University Hospital /ID# 164172, Vilnius
- Malaysia (4):
  - Hospital Sultanah Bahiyah /ID# 152310, Alor Star, Kedah
  - Hospital Ampang /ID# 152311, Ampang, Selangor
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 152313, Kuala Lumpur, Selangor
  - Uni Malaya MC /ID# 150440, Kuala Lumpur
- Mexico (3):
  - Morales Vargas Centro de Investigacion S.C. /ID# 211327, León, Guanajuato
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 202334, Guadalajara, Jalisco
  - Centro Regiomontano de Estudios Clínicos ROMA S.C /ID# 150265, Monterrey, Nuevo León
- Netherlands (5):
  - Radboud Universitair Medisch Centrum /ID# 151701, Nijmegen, Gelderland
  - Amsterdam UMC, locatie AMC /ID# 150617, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum /ID# 152625, Leiden, South Holland
  - Duplicate_Erasmus Medisch Centrum /ID# 150619, Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht /ID# 152776, Utrecht
- Norway (2):
  - Akershus Universitetssykehus_MAIN /ID# 150622, Lorenskog, Akershus
  - Universitetssykehuset I Nord-Norge /ID# 152836, Tromsø, Troms
- Poland (7):
  - Gastromed Sp. z o.o /ID# 216198, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Zdrowia MDM /ID# 150626, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 150627, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Reuma Park /ID# 150624, Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. /ID# 216743, Warsaw, Masovian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 215733, Warsaw, Masovian Voivodeship
  - Endoskopia Sp. z o.o. /ID# 152940, Sopot, Pomeranian Voivodeship
- Portugal (8):
  - Duplicate_Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 151616, Guimarães, Braga District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 152336, Santa Maria DA Feira, Porto District
  - Duplicate_Hospital Garcia de Orta, EPE /ID# 151622, Almada, Setúbal District
  - 2CA-Braga, Hospital de Braga /ID# 151617, Braga
  - Duplicate_Centro Hospitalar Universitario Lisboa Central, EPE - Hospital dos Cap /ID# 151620, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 151615, Lisbon
  - Unidade Local de Saude Sao Joao, EPE /ID# 151619, Porto
  - Unidade Local de Saude do Alto Minho, EPE /ID# 151618, Viana do Castelo
- School of Medicine University of Puerto Rico-Medical Science Campus /ID# 150629, San Juan, Puerto Rico
- Russia (10):
  - Immanuel Kant Baltic Federal University /ID# 202129, Kaliningrad, Kaliningrad Oblast
  - NW State Medical Univ na Mechn /ID# 169332, Saint Petersburg, Leningradskaya Oblast'
  - Republican hospital named after V.A. Baranov /ID# 206508, Petrozavodsk, Murmansk Oblast
  - Perm Clinical Center of the Federal Medical and Biological Agency /ID# 150634, Perm, Permskiy Kray
  - Medical Company Hepatology /ID# 200208, Samara, Samara Oblast
  - LLC Novaya Klinika /ID# 208106, Pyatigorsk, Stavropol Kray
  - Kazan State Medical University /ID# 166040, Kazan', Tatarstan, Respublika
  - Olla-Med Clinic /ID# 215334, Moscow
  - Euromedservice /ID# 208968, Pushkin
  - Duplicate_Stavropol State Medical Univ /ID# 150635, Stavropol
- Serbia (8):
  - Clinical Hosp Center Zvezdara /ID# 150641, Belgrade, Beograd
  - Military Medical Academy /ID# 150643, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 150642, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 150640, Belgrade, Beograd
  - General Hospital Leskovac /ID# 217882, Leskovac, Jablanicki Okrug
  - Duplicate_University Clinical Center of Nis /ID# 151902, Niš, Nisavski Okrug
  - University Clinical Center Kragujevac /ID# 150644, Kragujevac, Sumadijski Okrug
  - University Clinical Center Vojvodina /ID# 150759, Novi Sad
- Singapore (3):
  - National University Hospital /ID# 150583, Singapore
  - Gleneagles Medical Centre /ID# 206020, Singapore
  - Tan Tock Seng Hospital /ID# 150646, Singapore
- Slovakia (6):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 150869, Banská Bystrica, Banská Bystrica Region
  - B+B MED, s.r.o. /ID# 150584, Košice, Košice Region
  - Fakultna nemocnica s poliklinikou Nove Zamky /ID# 211371, Nové Zámky, Nitra Region
  - Gastro I., s.r.o. /ID# 150585, Prešov, Presov
  - Medak s.r.o. /ID# 150550, Bratislava
  - Slovak Research Center Team Me /ID# 150240, Ilava
- South Africa (8):
  - MD Search /ID# 157524, Boksburg North, Gauteng
  - Clinresco Centers /ID# 163625, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre /ID# 214361, Johannesburg, Gauteng
  - Wits Clinical Research /ID# 150586, Johannesburg, Gauteng
  - Wits Clinical Research , Wits Health Consortium (PTY) Ltd /ID# 157730, Johannesburg, Gauteng
  - Kingsbury Hospital /ID# 150587, Cape Town, Western Cape
  - Private Practice Dr MN Rajabally /ID# 155145, Cape Town, Western Cape
  - Spoke Research Inc /ID# 162203, CAPE TOWN Milnerton, Western Cape
- South Korea (10):
  - Dong-A University Medical Center /ID# 161568, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 161569, Busan, Busan Gwang Yeogsi
  - Duplicate_Hanyang University Gurihospital /ID# 150431, Guri-si, Gyeonggido
  - Duplicate_CHA University Bundang Medical Center /ID# 161567, Seongnam, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 150434, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 150435, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 159155, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 150433, Seoul, Seoul Teugbyeolsi
  - Yeungnam University Medical Center /ID# 150432, Daegu
  - Yonsei University Health System Severance Hospital /ID# 161566, Seoul
- Spain (10):
  - Complejo Hospitalario Universitario A Coruña /ID# 203912, A Coruña, A Coruna
  - Duplicate_Hospital Clínico Universitario de Santiago-CHUS /ID# 171492, Santiago de Compostela, A Coruna
  - Hospital Universitario Marques de Valdecilla /ID# 216621, Santander, Cantabria
  - Hospital Universitario Dr. Negrin /ID# 203965, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clinic de Barcelona /ID# 150598, Barcelona
  - Duplicate_Hospital Universitario Reina Sofia /ID# 154031, Córdoba
  - Hospital Universitario Ramon y Cajal /ID# 171491, Madrid
  - Hospital Universitario La Paz /ID# 214541, Madrid
  - Hospital Universitario de Salamanca /ID# 150590, Salamanca
  - Hospital Universitario y Politecnico La Fe /ID# 150591, Valencia
- Duplicate_Sahlgrenska University Hospital /ID# 152326, Gothenburg, Västra Götaland County, Sweden
- Switzerland (4):
  - University Hospital Basel /ID# 161732, Basel Town, Canton of Basel-City
  - Kantonsspital St. Gallen /ID# 152601, Sankt Gallen, Canton of St. Gallen
  - University Hospital Zurich /ID# 152603, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 152602, Bern
- Taiwan (6):
  - National Taiwan University Hospital /ID# 150604, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 150606, Kaohsiung City
  - Duplicate_Chung Shan Medical University Hospital /ID# 150603, Taichung
  - China Medical University Hospital /ID# 150600, Taichung
  - National Cheng Kung University Hospital /ID# 151751, Tainan
  - Taipei Veterans General Hosp /ID# 151750, Taipei
- Turkey (Türkiye) (6):
  - Gazi Universitesi Tip Fakultes /ID# 150493, Yenimahalle, Ankara
  - Duplicate_Erciyes University Medical Fac /ID# 150495, Melikgazi, Kayseri
  - Istanbul University Cerrahpasa Faculty of Medicine /ID# 150491, Cerrahpaşa
  - Umraniye Training and Res Hosp /ID# 163136, Istanbul
  - Marmara University Medical Fac /ID# 214573, Istanbul
  - Mersin University Medical /ID# 163135, Mersin
- Ukraine (10):
  - CNCE of Kharkiv Regional Council Regional Clinical Hospital /ID# 206941, Kharkiv, Kharkivs’ka Oblast’
  - Lviv Regional Clinical Hospital /ID# 150508, Lviv, Lviv Oblast
  - Municipal Non-Commercial Enterprise Odesa Regional Clinical Hospital of the Od /ID# 162502, Odesa, Odesa Oblast
  - Medical Center of the â€œHealth /ID# 162501, Vinnytsia, Vinnytsia Oblast
  - MNE Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 216302, Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "I.I. Mechnikov Dnipropetrovsk Regional Clinical Hospital" /ID# 207731, Dnipro
  - PE PMC Acinus, Medical and Diagnostic Center /ID# 217219, Kropyvnytskyi
  - Kyiv City Clinical Hospital No.18 /ID# 150505, Kyiv
  - Medical Center of LLC "Medical Center "Consilium Medical" /ID# 217448, Kyiv
  - CNPE of Kyiv Regional Council Kyiv Regional Hospital /ID# 217374, Kyiv
- United Kingdom (8):
  - Duplicate_Royal United Hospitals Bath /ID# 154211, Bath, Bath And North East Somerset
  - Royal Devon & Exeter Hospital /ID# 150510, Exeter, Devon
  - Hampshire Hospitals NHS Foundation Trust /ID# 150511, Basingstoke, Essex
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 150515, London, Greater London
  - Duplicate_St George's University Hospitals NHS Foundation Trust /ID# 208376, London, Greater London
  - Queen Elizabeth University Hospital - NHS Greater Glasgow and Clyde /ID# 163788, Glasgow, Lanarkshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 150513, Birmingham
  - Calderdale and Huddersfield NHS Foundation Trust /ID# 217659, Huddersfield

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Panaccione R, Vermeire S, Danese S, Higgins PDR, Lichtenstein GR, Nakase H, Glover S, Colombel JF, Eccleston J, Kujawski M, Remple V, Yao X, Geng Z, Palac H, Sharma D, Suravaram S, Schreiber S. Long-term efficacy and safety of upadacitinib in patients with moderately to severely active ulcerative colitis: an interim analysis of the phase 3 U-ACTIVATE long-term extension study. Lancet Gastroenterol Hepatol. 2025 Jun;10(6):507-519. doi: 10.1016/S2468-1253(25)00017-2. PMID 40347957
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/